CLINICAL TRIAL: NCT01479790
Title: Repeatability and Agreement of Visante and Cirrus Anterior Segment Optical Coherence Tomography and Functional Infrared Thermography
Brief Title: Repeatability and Agreement of Anterior Segment Optical Coherence Tomography (AS-OCT) and Thermography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Singapore Eye Research Institute (Other); Nanchang University (Other)
Responsible Party: Principal Investigator, Louis Tong, Clinician-Scientist, Consultant, Singapore National Eye Centre
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: R845/40/2011; 2011/408/A (Other: SingHealth Centralised Institutional Review Board)
Record Dates: First submitted 2011-10-04; First posted 2011-11-24 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Dry Eye Syndromes
Keywords: Visante AS-OCT; Cirrus AS-OCT; Thermography; Tear evaporation; Tear evaporimetry
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Visante AS-OCT and Cirrus AS-OCT (No Intervention): The tear meniscus is the thin concave strip of the tear film near the eyelid margins. During the acquisition the participants place their chins on a chin rest and look at a fixation light/target. This whole procedure should not take more than 5 minutes. The patients are allowed to blink freely except for during the acquisition time of less than 5 seconds. The procedure will be repeated for the upper and lower tear meniscus of both eyes.
- Thermography measurement (Experimental): In total, four pairs of thermographic sequences on the ocluar surface temperature from volunteers will be taken.
  1. A thermographic sequence will be captured from each eye.
  2. After 20 minutes, a second pair of thermographic sequences will be captured.
  3. An eye mask with a temperature of not more than 40 deg C (will be worn by the volunteer for 5 minutes and a third pair of thermographic sequences will be captured immediately after mask removal.
  4. A fourth pair of thermographic sequences will be captured 1 hour after mask removal.
  Interventions: Device: EyeGiene

INTERVENTIONS:
Device: EyeGiene — The eye mask with a temperature of not more than 40 deg C (confirmed by thermometer) will be worn by the volunteer for 5 minutes.
  Other Names: EyeGiene (Eyedetec Medical Inc., US)
  Arms: Thermography measurement

SUMMARY:
Dry eye is a common condition that affects vision and quality of life in patients. Dry eye clinical research is limited to follow up of disease progression. Currently, most research outcomes are based on subjective patient complaints rather than objective assessment of the condition. Only few objective measurements for dry eye are available today and this is mainly the result of poor repeatability and inaccuracy.

This current study aims to evaluate 2 new non-invasive imaging techniques suitable for dry eye assessment.

Anterior segment optical coherence tomography (AS-OCT) is an imaging device that has the ability to image the tear meniscus of the eye in a safe and non-invasive manner. Image analysis can then indirectly determine the tear film volume. Improvements in the image resolution of these devices require a study that compares the repeatability and agreement of an older (Visante AS-OCT) and a newer instrument (Cirrus AS-OCT) which the current study aims to address.

Another method of evaluating dry eye disease is a novel technique that uses functional infrared thermography to measure tear evaporation rate. This study will also establish repeatability of measurements of the ocular surface temperature which are used to calculate tear evaporation rates.

Should these methods are found to be repeatable, they can be used in future clinical trials as an additional tool to investigate dry eye treatments.

DETAILED DESCRIPTION:
Study Objectives and Purpose:

Part A - AS-OCT repeatability and agreement

1. The primary purpose of Part A is to compare the repeatability of the Cirrus with the Visante AS-OCT imaging system.
2. The second objective is to identify the level of agreement in the tear meniscus measurements taken by the Cirrus and Visante AS-OCT.

Part B - Tear evaporimetry with functional infra-red thermography

1. To evaluate the repeatability of Infrared thermography for ocular surface temperature measurements that are used for calculation of tear evaporation rates. If this is found to be acceptable, it will be correlated to tear meniscus parameters.
2. To determine whether this method is able to detect temperature changes of the ocular surface.

Study design:

Part A. Cross sectional study. Part B. Prospective study

Rationale:

Part A - AS-OCT repeatability and agreement Repeatability is an important issue in the objective assessment of dry eye. While previous studies have compared various methods of measuring the tear meniscus, including the use of Visante AS-OCT, current literature lacks studies that investigated the Cirrus AS-OCT for assessment of dry eye. With a higher resolution, the Cirrus is potentially useful as a non-invasive procedure for objective measurements of the tear meniscus.

Part B - Tear evaporimetry with functional infra-red thermography Current available methods to measure of tear evaporation rate have major limitations. This new method, however, is non-invasive, has no need for special eye drops or chambers and takes temperature measurements very quickly. This method is therefore extremely practical and provides many exciting possibilities for future trials.

Methods:

Participants and target sample size 40 volunteers from Singapore Eye Research Institute will be recruited for this study. Each volunteer will be given a study serial number to ensure anonymity.

20 will participate in the AS-OCT study. 20 will participate in the tear evaporimetry study.

Part A - AS-OCT repeatability and agreement Two AS-OCT imaging systems, namely Cirrus and the Visante, will be tested. All participants undergo acquisition of 2 images by the Visante AS-OCT, then 2 images by the Cirrus AS-OCT. Both images will be acquired by the same technician.

Part B - Tear evaporimetry with functional infra-red thermography In total, four pairs of thermographic sequences on the ocluar surface temperature from volunteers will be taken.

1. The volunteer will be seated in front of the thermographic camera and on each eye on thermographic sequence will be captured.
2. After 20 minutes, a second pair of thermographic sequences will be captured.
3. An eye mask with a temperature of not more than 40 deg C (confirmed by thermometer) will be worn by the volunteer for 5 minutes.
4. A third pair of thermographic sequences will be captured immediately after mask removal.
5. A fourth pair of thermographic sequences will be captured 1 hour after mask removal.

Between sequence acquisitions, the volunteer is allowed to move freely in the room. The temperature and humidity of the room will be kept constant during measurements.

Visit schedules:

Only one examination per ASOCT instrument for Part A is required. For Part B, all thermography will be performed on the same day.

If participants agree to have both ASOCT and tear evaporimetry done, then they will undergo Parts A and B. If not, they will be recruited for either Part A or Part B.

Duration of study: 1 day

ELIGIBILITY:
Inclusion Criteria:

- Volunteers that are medically fit and willing to participate in this study.

Exclusion Criteria:

* No eye surgery done within the previous 3 months
* Active ocular infection or pterygium that may affect tear film stability.
* Any other specified reason as determined by clinical investigator.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
equipment repeatability | 1 day
  Part A - The repeatabilty coefficients of tear meniscus measurements derived from Visante and Cirrus AS-OCT and the agreement between tear meniscus measurements.
  Part B - Infrared thermography is expected to be repeatable in capturing OST measurements which will consequently result in repeatable tear evaporation rates. Temperature changes of the ocular surface will be adequately captured.

SECONDARY OUTCOMES:
temperature changes | 1 day
  Determine whether thermogram images can capture changes in temperature/the rate of tear evaporation which were introduced by warm eye mask wear.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Tong, PhD, Principal Investigator — Singapore National Eye Centre
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore, Singapore

REFERENCES:
- [Background] Tan JH, Ng EY, Acharya UR. Evaluation of tear evaporation from ocular surface by functional infrared thermography. Med Phys. 2010 Nov;37(11):6022-34. doi: 10.1118/1.3495540. PMID 21158314
- [Background] Savini G, Goto E, Carbonelli M, Barboni P, Huang D. Agreement between stratus and visante optical coherence tomography systems in tear meniscus measurements. Cornea. 2009 Feb;28(2):148-51. doi: 10.1097/ICO.0b013e31818526d0. PMID 19158555